CLINICAL TRIAL: NCT06972537
Title: Model-Guided Dose Optimization vs. Empirical Dosing of Piperacillin-Tazobactam in the Treatment of Pneumonia in Elderly Patients: A Study on Superiority
Brief Title: A Study on the Infusion Regimen of Piperacillin-Tazobactam in Patients Aged 65 and Older With Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SDU-2024-PIP-002
Record Dates: First submitted 2025-04-16; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Tazobactam; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empirical regimen (Active Comparator): Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda) 4.5g, administered every 8 hours, with each infusion lasting for 3 hours
  Interventions: Drug: Extended Infusion Time of Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda), 4.5g
- Prolonged infusion time (Experimental): Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda) 4.5g, administered every 6 hours, with each infusion lasting for 4 hours
  Interventions: Drug: Increase the frequency and extended infusion time of Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda) 4.5g

INTERVENTIONS:
Drug: Increase the frequency and extended infusion time of Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda) 4.5g — Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda) 4.5g administered four times a day (QID), with each infusion lasting for 4 hours.
  Arms: Prolonged infusion time
Drug: Extended Infusion Time of Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda), 4.5g — Piperacillin Sodium and Tazobactam Sodium for Injection (Bonda), 4.5g administered three times a day (TID), with each infusion lasting for 3 hours.
  Arms: Empirical regimen

SUMMARY:
Pneumonia is characterized by high incidence and mortality rates in elderly patients (≥65 years old). Piperacillin-tazobactam, as a broad-spectrum antibiotic, has its therapeutic efficacy and safety potentially influenced by the infusion regimen. However, research on infusion regimens specifically targeting the elderly population is currently limited. In our preliminary dose simulation, under the pharmacokinetic/pharmacodynamic (PK/PD) target of achieving a free drug concentration time percentage above 100% of the minimum inhibitory concentration (fT%>100% MIC), the regimen of administering the drug every 6 hours (q6h) achieved a concentration compliance rate of 90% within 4 hours. This study aims to explore the differences between two infusion modes (q6h for 4 hours vs. q8h for 3 hours) and to provide preliminary evidence for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Age must be greater than 65 years Clinical diagnosis of Pneumonia Receiving intravenous piperacillin-tazobactam treatment

Exclusion Criteria:

History of allergy to β-lactam antibiotics Continuous renal replacement therapy, severe organ dysfunction Malignant tumor disease

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement rate | 3 months
  Improvement in pneumonia symptoms, such as normalization of body temperature (temperature reduced to 37.8°C or below and maintained for 48 hours), alleviation of symptoms (coughing subsides, sputum production decreases, dyspnea eases, respiratory rate drops to below 24 breaths per minute, and other symptoms such as fatigue and chest pain significantly improve), improvement in physical signs (heart rate decreases to below 100 beats per minute, and wet rales on lung auscultation diminish or disappear), improvement in laboratory tests (white blood cell count returns to normal or near-normal levels, and levels of inflammatory markers such as C-reactive protein and procalcitonin decline), and radiological improvement (chest X-ray or CT shows absorption of pulmonary inflammation and reduction in the extent of lesions), as well as the Apache II score.

SECONDARY OUTCOMES:
PK/PD target attainment rate | 2 days
28-day mortality rate | 3 months
7-day microbiological clearance rate | after 7days when finished infuse piperacillin
Length of Hospital Stay ICU and Length of ICU Stay | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Second hospital of Shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes